CLINICAL TRIAL: NCT05308485
Title: Events Exposure as a Trigger of the Clinical Manifestations of Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fundación para la Lucha contra las Enfermedades Neurológicas de la Infancia (Other)
Responsible Party: Principal Investigator, Malco Rossi, MD, PhD - Co-investigator - Clinical Professor, Fundación para la Lucha contra las Enfermedades Neurológicas de la Infancia
Other Study IDs: 3961
Record Dates: First submitted 2022-03-24; First posted 2022-04-04 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-03

CONDITIONS: Parkinson Disease; Parkinsonism
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Parkinson´s disease individuals
  Interventions: Other: Events exposure questionnaire
- Individuals with recent-onset parkinsonism
  Interventions: Other: Events exposure questionnaire
- Healthy individuals
  Interventions: Other: Events exposure questionnaire

INTERVENTIONS:
Other: Events exposure questionnaire — Events exposure questionnaire that assess the occurrence of exposure to events and their severity over a limited period

SUMMARY:
Stress has been implicated as a trigger of many diseases, throughout different mechanisms. Potentially traumatic/stressful events exposure might be a factor that triggers subclinical disabilities related to PD becoming evident to the patient. In this observational study, the investigators will evaluate with a validated events exposure questionnaire the occurrence and severity of potentially traumatic or stressful events in Parkinson's disease patients and in patients with recent-onset parkinsonism.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is one of the most common neurodegenerative disorders worldwide, affecting approximately 1% of individuals older than 60 years and causing progressive disability. Clinical signs and symptoms of PD include asymmetric bradykinesia, rest tremor, rigidity, postural instability, and gait abnormalities.

Stress has been implicated as a trigger of many diseases, throughout different mechanisms. Potentially traumatic/stressful events exposure might be a factor that triggers subclinical disabilities related to PD becoming evident to the patient. Stress or events exposure can be associated with the clinical expression of Parkinson's sisease, acting as the final hit in a predisposed person. The prevalence of exposure to traumatic events (TE) throughout life in different populations has been analyzed in multiple studies, with variable percentages, ranging from 30 -70%.

It is well known that stress activates both the sympathetic nervous system and the hypothalamic - pituitary - adrenal (HPA) axis, resulting in increases in the secretion of catecholamines and glucocorticoids (GCs) into the peripheral circulation. Stress also can increase the release of dopamine (DA) and glutamate in the striatum as well as other brain regions. It is likely that these effects of stress have evolved as part of a generalized response to potential danger, facilitating the ability of the organism to respond appropriately to the stressor. More specifically, given the impact of DA and glutamate on striatal function, these changes can be expected to increase the capacity of the CNS to focus, process, and ultimately respond appropriately to emergencies. These effects are likely to be reinforced by the increased availability of GCs. Yet, when the amplitude or duration of these biological changes becomes excessive, the possibility of neuronal cell death develops. The greatest risk factor for PD appears to be age. The tendency for the symptoms of PD to emerge after the age of 55 may be due in part to a failure of compensatory mechanisms that underlie the extended preclinical phase of the disease. However, it is likely that another factor in the late onset of PD is the increased vulnerability of DA neurons to insult. In this regard, it is important to note that dysfunctions in the stress response develop during the aging process. For example, as organism ages, the response of the HPA axis to stress becomes hyperactive and is slower to return to homeostatic conditions after activation, thus exposing cells to higher levels of GCs for a prolonged period. This dysregulation might render cells in the aged brain more susceptible to degeneration in the face of subsequent stress.

In this observational study, the investigators will evaluate with a validated events exposure questionnaire the occurrence and severity of potentially traumatic or stressful events in Parkinson's disease patients and in patients with recent-onset parkinsonism.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent is obtained from the participant
* The participant is clinically diagnosed with Parkinson's disease
* The participant has recent-onset parkinsonism

Exclusion Criteria:

* Participants with parkinsonism with more than 4 years of evolution of the disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinically diagnosed Parkinson's Disease (PD) patients and patients with recent-onset parkinsonism
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2022-07-26 (Estimated); Study Completion 2022-07-27 (Estimated)

PRIMARY OUTCOMES:
Recruitment of 300 participants | 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- FLENI, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: No
The plan will be defined at a later stages

REFERENCES:
- [Result] Paez-Maggio M, Rossi M, Fazzito L, Merello M. Validation of an events exposure questionnaire for individuals living in major cities of Argentina. Eur J Psychotraumatol. 2022 Feb 15;13(1):2031830. doi: 10.1080/20008198.2022.2031830. eCollection 2022. PMID 35186218